CLINICAL TRIAL: NCT01948895
Title: An 8-week Open-Label Flexible-Dose Study Of Desvenlafaxine as Monotherapy In The Treatment Of Dysthymia
Brief Title: Desvenlafaxine Monotherapy in Dysthymia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Principal Investigator, Arun Ravindran, Principal Investigator, Centre for Addiction and Mental Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 124/2012
Record Dates: First submitted 2013-09-19; First posted 2013-09-24 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Dysthymic Disorder
Keywords: Desvenlafaxine; Open-label; Flexible-dose; Dysthymic disorder; Anxiety disorders; Generalized anxiety disorder; Social anxiety disorder; Post-traumatic stress disorder
MeSH Terms: conditions — Dysthymic Disorder; Anxiety Disorders; Generalized Anxiety Disorder; Phobia, Social; Stress Disorders, Post-Traumatic | interventions — Desvenlafaxine Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single-arm study (Experimental): Desvenlafaxine 50mg/day Desvenlafaxine 100mg/day
  Interventions: Drug: Desvenlafaxine

INTERVENTIONS:
Drug: Desvenlafaxine — Patients will be initiated on 50 mg/day of Desvenlafaxine. No dose changes will be allowed for the first four weeks. If there is partial or no response after four weeks, dosage will then be increased to 100mg/day, based on tolerability and the Investigator's judgment.
  Other Names: Pristiq

SUMMARY:
This multi-centred study will be conducted at two centres. The design will be an open label, flexible-dose study. This investigation will evaluate the efficacy of Desvenlafaxine monotherapy for patients who meet diagnostic criteria for dysthymia.

DETAILED DESCRIPTION:
Primary objective: To investigate the efficacy, safety, and tolerability of open-label desvenlafaxine monotherapy in dysthymic subjects.

Secondary objectives: To evaluate the efficacy of desvenlafaxine on clinical measures relating to improvement of depressive symptoms, quality of life and occupational functioning.

It is hypothesized that Dysthymic subjects will show significant improvement in depressive symptoms after 8 weeks of treatment with desvenlafaxine. There will be significant improvement in measures of quality of life and stress coping at end of treatment, compared to Baseline. There will also be significant improvement in measures of occupational functioning at end of treatment, compared to Baseline.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients between 18-65 years.
* Primary diagnosis of Dysthymic Disorder, as defined by DSM-IV criteria (300.4).
* MADRS score ≥15 at Screening and Baseline.
* Supportive therapy, and use of zopiclone for sleep and low-dose benzodiazepines on an as needed basis for anxiety, is allowed at any time.
* Written informed consent

Exclusion Criteria:

* Co-morbid diagnosis of any other Axis I disorders (other than anxiety disorders such as Generalized Anxiety Disorder, Social Anxiety Disorder and Post-traumatic Stress Disorder, provided that Dysthymic Disorder is currently the diagnosis).
* Meet DSM-IV criteria for a current episode of major depression within two months prior to screening or who have received treatment for a major depressive episode within six months prior to screening.
* Substance abuse or dependence including alcohol, within 6 months prior to screening.
* Patients on the following prohibited treatments:

  1. Psychotropics such as other SSRIs, other SNRIs, lithium, sibutramine, tramadol, St. John's Wort, within 2 weeks of randomization
  2. Agents that impact significantly on serotonin metabolism (e.g. MAOIs, tryptophan, triptans) within 2 weeks of randomization
* Have received physical therapies for depression (e.g. ECT, rTMS) within the 3 months prior to randomization.
* Previous non-response to a therapeutic trial of desvenlafaxine (at least 50 mg/day for 2 months).
* Clinically significant abnormalities in hematology, clinical chemistry, urinalysis or ECG at the screening visit, as judged by the Principal Investigator.
* Presence of medical or psychiatric condition deemed by the Investigator to interfere with study procedures or endpoint data.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Montgomery-Åsberg Depression Rating Scale | 8 Weeks

SECONDARY OUTCOMES:
Clinical Global Impression Scale | 8 Weeks
Health and Work Performance Questionnaire | Baseline, Week 8
Perceived Stress Scale | Baseline, Week 8
Quality of Life Enjoyment and Satisfaction Scale Quality of Life Enjoyment and Satisfaction Scale Quality of Life Enjoyment and Satisfaction Questionnaire | Baseline, Week 4, Week 8
Quick Inventory of Depressive Symptomatology | Baseline, Week 4, Week 8
Survey of Coping Profiles Endorsed | Baseline, Week 4, Week 8
Sheehan Disability Scale | Baseline, Week 4, Week 8
Work Productivity and Activity Impairment Questionnaire | Baseline, Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Arun Ravindran, MD, PhD, Principal Investigator — Centre for Addiction and Mental Health
Locations (2):
- Canada (2):
  - Medical Research Associates, Mississauga, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario

REFERENCES:
- See also: Information about research at the Centre for Addiction and Mental Health — http://www.camh.ca/en/research/Pages/research.aspx